CLINICAL TRIAL: NCT06519942
Title: Muscle and Bone in Patients with Diabetes Mellitus and Neuropathy
Acronym: SVT-DNP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0120; BOF.24Y.2023.0030.01 (Other Grant/Funding Number: Special Research Fund (Ghent University))
Record Dates: First submitted 2024-04-10; First posted 2024-07-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Peripheral Neuropathy; Sarcopenia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sarcopenia | interventions — Blood Specimen Collection; Electrocardiography; Surveys and Questionnaires; Anthropometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood sample, muscle biopsy sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- T2DM DNP+: type 2 diabetes with diabetic neuropathy
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Electromyoneurography (EMNG); Procedure: Muscle biopsy; Radiation: Quantitative peripheral computed tomography (qPCT); Device: Mechanography; Diagnostic Test: Electrocardiography (ECG); Other: Questionnaires; Other: Anthropometry
- T2DM DNP-: type 2 diabetes without diabetic neuropathy
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Electromyoneurography (EMNG); Procedure: Muscle biopsy; Radiation: Quantitative peripheral computed tomography (qPCT); Device: Mechanography; Diagnostic Test: Electrocardiography (ECG); Other: Questionnaires; Other: Anthropometry
- HC: healthy controls
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Electromyoneurography (EMNG); Procedure: Muscle biopsy; Radiation: Quantitative peripheral computed tomography (qPCT); Device: Mechanography; Diagnostic Test: Electrocardiography (ECG); Other: Questionnaires; Other: Anthropometry

INTERVENTIONS:
Diagnostic Test: Blood sampling — Fasting blood samples will be obtained.
Diagnostic Test: Electromyoneurography (EMNG) — Nerve conduction of sensory and motor nerves of the upper and lower limb will be performed, including F- and H-waves. Needle EMNG of the m. tibialis anterior, m. gastrocnemius (medial head), m. tensor fascia lata and m. gluteus maximus) will be performed.
Procedure: Muscle biopsy — Muscle biopsy of the m. gastrocnemius will be performed under local anesthesia using the modified Bergström technique.
Radiation: Quantitative peripheral computed tomography (qPCT) — A qPCT scan of the calf will be performed.
Device: Mechanography — Single two leg jump, multiple one leg hopping, chair rise and sit to stand tests will be performed.
Diagnostic Test: Electrocardiography (ECG) — A 15-minute resting ECG will be performed.
Other: Questionnaires — Questionnaires will be performed to collect information on medical background (drug use, comorbidities, symptoms of peripheral neuropathy, ...) and lifestyle factors (ethyl consumption, food intake, physical activity, smoking).
Other: Anthropometry — Length and hip:waist ratio will be measured. Furthermore, body weight and composition will be determined by bio-impedance measurement. Systolic and diastolic blood pressure (mean of 3 times) will be evaluated.

SUMMARY:
The goal of this observational study is to evaluate muscle fiber type composition in people with type 2 diabetes mellitus (T2DM) with a common complication of T2DM: diabetic peripheral neuropathy (DNP), specifically diabetic sensorimotor polyneuropathy. Researchers will also look into factors related to DNP: inflammation, the use of energy in the cell, nerve function and the tiny blood vessels in the muscle.

The main question it aims to answer is: Are there differences in muscle fiber type composition between persons with T2DM with and without DNP, in comparison to sex and age-matched healthy peers?

Participants will partake in the following tests:

* electromyoneurography (EMNG): evaluation of nerve function, damage and repair; for diagnosis of DNP or other diseases of the nerves
* blood analysis: researchers will measure insulin, blood sugar, lipid profile, inflammation
* muscle biopsy in the calf (m. gastrocnemius): a doctor will take a small sample of muscle to evaluate the muscle shape and structure
* mechanography: patients will perform functional tests (e.g. standing up from a chair), researchers will evaluate maximal power and maximal force of the muscles by jumping tests
* questionnaires: on food intake, physical activity, smoking history, alcohol use, medical history
* measurement of height, weight, and the comparison of the hip and waist circumference
* peripheral Quantitative Computed Tomography (pQCT): scan of the calf for muscle density and bone density
* electrocardiography (ECG): evaluation of electrical signals of the heart

Researchers will compare (1) patients with T2DM with DNP, (2) patients with T2DM without DNP, and (3) healthy persons to see if there are differences in muscle fiber type composition

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Between 40-70 years of age
* BMI between 18,5 - 35 kg/m2

Persons with T2DM:

* More than 10-year clinical diagnosis of T2DM

Exclusion Criteria:

All participants:

* Possible other causes of nerve impairment (vitamin B12 deficiency, excessive alcohol consumption, chemotherapy)
* Immobilisation (1) > 3 months in past history or (2) > 4 weeks in past 6 months
* Chronic conditions affecting the vital organs (New York Heart Association (NYHA) 3/4, Global Initiative for Obstructive Lung Disease (GOLD) 3/4, cystic fibrosis)
* Hypogonadism
* Inflammatory joint or intestinal diseases
* Chronic muscle diseases
* Active malignancy
* Malnutrition disease, eating disorder or bariatric surgery
* Medication use (anticoagulants, glucocorticoids, anti-androgen or anti-estrogen treatment) persons with T2DM:
* Insufficient control of diabetes (HbA1c >9%)

Healthy controls:

* Fasting glucose > 100 mg/dl
* HbA1c > 5.7 %

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited through the Ghent University Hospital, diabetes educators and podologists.
Sampling Method: Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Differences in muscle fiber type composition in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Differences in muscle fiber type distribution, percentage and cross-sectional area will be evaluated through myosin heavy chain (MHC) immunostaining of the muscle specimen.

SECONDARY OUTCOMES:
Differences in nerve conduction velocity in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls | At enrollment
  Nerve conduction velocity will be examined through EMNG examination to examine neuromotor function
Differences in capillarization in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Capillarization will be examined through histological examination of the muscle specimen using Ulex europaeus I (UEA-I) staining.
Differences in electron microscopic properties assessing mitochondrial function in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls | At enrollment
  Mitochondrial function will be examined through electron microscopy of the muscle specimen.
Differences in maximal force in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Maximal force will be evaluated using mechanography through multiple one leg hopping.
Differences in maximal power in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Maximal power will be evaluated using mechanography through the single two leg jump.
Differences in functional muscle strength in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Functional strength will be examined using mechanography through the chair rising test and heel rise test.
Differences in physical activity levels in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Differences in the lifestyle factor physical activity will be examined through the International Physical Activity Questionnaire (IPAQ) - Long Form).
Differences in food intake in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Differences in the lifestyle factor food intake will be examined through a food frequency questionnaire.
Differences in lifestyle factors in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Differences in lifestyle factors smoking and ethyl consumption will be examined through non-official questionnaires.
Differences in muscle density in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Differences in muscle density will be evaluated through pQCT of the calf.
Differences in bone density in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Differences in bone density will be evaluated through pQCT of the calf.

OTHER OUTCOMES:
Differences in heart rate variability in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Heart rate variability will be examined through a 15-minute resting ECG.
Differences in interleukin 6 (IL-6) concentration in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Differences in inflammation will be evaluated through blood analysis of IL-6.
Differences in tumor necrosis factor alpha (TNFα) concentration in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Differences in inflammation will be evaluated through blood analysis of TNFα.
Differences in C-reactive protein (CRP) concentration in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Differences in inflammation will be evaluated through blood analysis of CRP.
Differences in mononuclear cell numbers in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Differences in inflammation will be evaluated through flow cytometry to assess mononuclear cell numbers.
Differences in protein concentrations for AMPK and PGC-1α in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls | At enrollment
  Differences in protein concentrations for 5' adenosine monophosphate-activated protein kinase (AMPK) and peroxisome proliferator-activated receptor-gamma coactivator 1 alpha (PGC-1α) will be examined using western blotting (on the muscle sample)
Differences in citrate synthase activity in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls | At enrollment
  Citrate synthase activity will be examined using an activity assay (on the muscle sample).
Differences in succinate dehydrogenase B (SDHB) expression in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls | At enrollment
  SDHB expression will be examined through immunohistochemical staining for SDHB of the muscle specimen.
Differences in vascular endothelial growth factor (VEGF) concentrations in persons with type 2 diabetes with diabetic peripheral neuropathy compared to persons with type 2 diabetes without diabetic neuropathy and healthy controls. | At enrollment
  Vascular endothelial growth factor concentrations will be examined through blood analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Lapauw, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
After publication, anonymous individual participant data can be made available to other researchers upon request.
Supporting Information: Study Protocol, ICF
Time Frame: After publication
Access Criteria: Upon request to corresponding author